CLINICAL TRIAL: NCT02330328
Title: Evaluation of the Utility of Telemetry in Patients Admitted for Chest Pain Who Are at Low Risk for Acute Coronary Syndrome
Brief Title: Telemetry for Chest Pain of Low Risk for Acute Coronary Syndrome Pts
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Collaborator withdrew closing the study prematurely with no participants enrolled
Sponsor: Carilion Clinic (Other)
Collaborators: Johns Hopkins University (Other); University of Maryland, College Park (Other); Virginia Commonwealth University (Other); Medstar Health Research Institute (Other); Virginia Tech Carilion School of Medicine and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NA_00091964
Record Dates: First submitted 2014-12-31; First posted 2015-01-01 (Estimated); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Chest Pain; Telemetry; Acute Coronary Syndrome; Health Care Resource Utilization
Keywords: Chest Pain; Telemetry
MeSH Terms: conditions — Chest Pain; Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No Telemetry Monitoring (Experimental): The participants in this arm will be admitted to a bed without telemetry monitoring
  Interventions: Other: No Telemetry Monitoring
- Telemetry (Active Comparator): The participants in this arm will be admitted to a bed with telemetry monitoring
  Interventions: Device: Telemetry Monitoring

INTERVENTIONS:
Other: No Telemetry Monitoring
  Arms: No Telemetry Monitoring
Device: Telemetry Monitoring
  Arms: Telemetry

SUMMARY:
This is a randomized controlled, multi-center, non-blinded non-inferiority study examining the utility of telemetry monitoring in patients admitted who are low risk for acute coronary syndrome. Each of the six sites will prospectively enroll 250 patients in each arm of the study randomized to either a med-surg bed (no telemetry) or a telemetry bed during their admission. Research study coordinators will enroll patients and then follow them throughout their hospital course and record primary and secondary end point events.

DETAILED DESCRIPTION:
This is a randomized controlled, multi-center, non-blinded non-inferiority study examining the utility of telemetry monitoring in patients admitted who are low risk for acute coronary syndrome. Each of the six sites will prospectively enroll 250 patients in each arm of the study randomized to either a med-surg bed (no telemetry) or a telemetry bed during their admission. Research study coordinators will enroll patients and then follow them throughout their hospital course and record primary and secondary end point events.

The research coordinators will collect information on the following items for data collection: age, gender, smoking history, history of hypertension, history of diabetes mellitus, history of hypercholesterolemia, and history of family member with early heart disease or myocardial infarction, and body mass index. Research coordinators will document if the patient had any of the following events during their hospital course: death, myocardial infarction (MI), upgrade to a higher level of care, dysrhythmia, results of any stress testing or cardiac catheterization. In addition patients will be contacted at 30 days and 365 days to inquire about MI, needing for percutaneous coronary intervention (PCI), or revascularization (CABG).

Based on previous studies, we hypothesize that patients aged 18-49 years who are at low risk for Acute Coronary Syndrome (ACS) are unlikely to benefit from continuous heart monitoring while admitted to the hospital for chest pain. We suspect that the rate of significant events may approach zero in this group of participants. This study aim is to show that a bed without remote monitoring- telemetry- is adequate when these low risk participants with chest pain are hospitalized.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be admitted for chest pain and evaluation of acute coronary syndrome

Exclusion Criteria:

* History of coronary artery disease, previous myocardial infarction, or any percutaneous intervention either documented in the medical report or verbal report by patient
* Have an initial troponin serum value above the threshold for that hospital's normal limit
* Have used cocaine in the previous 14 days (patient report)
* Have an abnormal ECG as determined by attending emergency physician
* Unable to consent for the study due to language barrier or mental incapacity
* Admitting attending physician does not agree with randomization of the patient into either study arm
* Pregnancy

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Sustained (> 30 seconds) or symptomatic ventricular tachycardia | up to 60 sec
Ventricular fibrillation | Baseline
Death | up to 1 year after enrollment

SECONDARY OUTCOMES:
Non-ST Segment Elevation Myocardial Infarction (NSTEMI) | Baseline, 30 days and 1 year after enrollment
ST Segment Elevation Myocardial Infarction (STEMI) | Baseline, 30 days and 1 year from enrollment
Positive Stress Test | Baseline, 30 days and 1 year after enrollment
Negative Stress Test | Baseline, 30 days and 1 year after enrollment
Cardiac catheterization result | Baseline, 30 days and 1 year after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: John Perkins, MD, Principal Investigator — Carlion Clinic

REFERENCES:
- [Background] Estrada CA, Rosman HS, Prasad NK, Battilana G, Alexander M, Held AC, Young MJ. Role of telemetry monitoring in the non-intensive care unit. Am J Cardiol. 1995 Nov 1;76(12):960-5. doi: 10.1016/s0002-9149(99)80270-7. PMID 7484840
- [Background] Hollander JE, Sites FD, Pollack CV Jr, Shofer FS. Lack of utility of telemetry monitoring for identification of cardiac death and life-threatening ventricular dysrhythmias in low-risk patients with chest pain. Ann Emerg Med. 2004 Jan;43(1):71-6. doi: 10.1016/s0196-0644(03)00719-4. PMID 14707944
- [Background] Durairaj L, Reilly B, Das K, Smith C, Acob C, Husain S, Saquib M, Ganschow P, Evans A, McNutt R. Emergency department admissions to inpatient cardiac telemetry beds: a prospective cohort study of risk stratification and outcomes. Am J Med. 2001 Jan;110(1):7-11. doi: 10.1016/s0002-9343(00)00640-9. PMID 11152858
- [Background] O'Neill DR. Low-risk classified chest pain patients: Do they need cardiac monitoring in the emergency department and can they be cared for in non-monitored beds? Australian Emerg Nur J 2007; 10:58-63.
- [Background] Perkins JC, Voore N, Patel J, et al: Assessment of an Emergency Department Chest Pain Patient Cohort at Low Risk for Significant Adverse Events During Admission for Acute Coronary Syndrome. SAEM Mid-Atlantic Regional Meeting, 02/2014, Philadephia, PA.
- [Background] Perkins J, McCurdy MT, Vilke GM, Al-Marshad AA. Telemetry bed usage for patients with low-risk chest pain: review of the literature for the clinician. J Emerg Med. 2014 Feb;46(2):273-7. doi: 10.1016/j.jemermed.2013.08.098. Epub 2013 Nov 22. PMID 24268896
- [Background] Hermann LK, Weingart SD, Duvall WL, Henzlova MJ. The limited utility of routine cardiac stress testing in emergency department chest pain patients younger than 40 years. Ann Emerg Med. 2009 Jul;54(1):12-6. doi: 10.1016/j.annemergmed.2009.01.006. Epub 2009 Feb 23. PMID 19231025
- [Background] Collin MJ, Weisenthal B, Walsh KM, McCusker CM, Shofer FS, Hollander JE. Young patients with chest pain: 1-year outcomes. Am J Emerg Med. 2011 Mar;29(3):265-70. doi: 10.1016/j.ajem.2009.09.031. Epub 2010 Mar 25. PMID 20825795
- [Background] Than M, Cullen L, Aldous S, Parsonage WA, Reid CM, Greenslade J, Flaws D, Hammett CJ, Beam DM, Ardagh MW, Troughton R, Brown AF, George P, Florkowski CM, Kline JA, Peacock WF, Maisel AS, Lim SH, Lamanna A, Richards AM. 2-Hour accelerated diagnostic protocol to assess patients with chest pain symptoms using contemporary troponins as the only biomarker: the ADAPT trial. J Am Coll Cardiol. 2012 Jun 5;59(23):2091-8. doi: 10.1016/j.jacc.2012.02.035. Epub 2012 May 9. PMID 22578923
- [Background] Henriques-Forsythe MN, Ivonye CC, Jamched U, Kamuguisha LK, Olejeme KA, Onwuanyi AE. Is telemetry overused? Is it as helpful as thought? Cleve Clin J Med. 2009 Jun;76(6):368-72. doi: 10.3949/ccjm.76a.07260. PMID 19487558
- See also: Telemetry bed usage for patient with low risk chest pain. — http://www.aaem.org/UserFiles/file/4.11.11BODApprvdTelemetryWebPosting.pdf